CLINICAL TRIAL: NCT06323941
Title: Effects of Motor Imagery on Skin Conductance and Pelvic Floor Sensorimotor Condition in Healthy Women: A Randomized Controlled Trial
Brief Title: Motor Imagery and Isometric Exercises on Pelvic Floor Sensorimotor Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Ferran Cuenca, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UV0003
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Isometric Exercise; Motor Imagery; Women's Health
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery plus Isometric Exercise (Experimental): This group will perform a therapeutic exercise programme (isometric exercises training) to which motor imagery training will be added.
  Interventions: Behavioral: Motor Imagery plus therapeutic exercise
- Isometric Exercise (Active Comparator): This group will perform a therapeutic exercise programme (isometric exercises training) to which sham motor imagery training will be added.
  Interventions: Behavioral: Therapeutic exercises

INTERVENTIONS:
Behavioral: Motor Imagery plus therapeutic exercise — Isometric exercises (20 minutes) to which will be added a motor imagery intervention (imagining movements without actually doing them).
  Arms: Motor Imagery plus Isometric Exercise
Behavioral: Therapeutic exercises — Isometric exercises (20 minutes) to which will be added a placebo motor imagery intervention (imagining a blue sky).
  Arms: Isometric Exercise

SUMMARY:
Mental practice (both in isolation and also in combination with real practice) has been shown to improve somatosensory and motor variables but so far no study has taken it into the study of women's health. Through the present study the investigators want to offer some interesting data regarding the effectiveness of mental practice combined with physical practice.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age and asymptomatic women.

Exclusion Criteria:

* This study will exclude those who presented a respiratory pathology, cardiac, systematic, or metabolic disease, history of recent surgery, vertebral fracture, or osteoarticular disorders of the spine area.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Skin conductance (for asessing electrodermal activity) | pre-intervention (T0), and inmmediate post-intervention (T1) (between the first and the second measurement, about 60 minutes have elapsed because it is done on the same day)
  skin conductance is a measure of sweating which is an excitatory sympathetic monoinervative variable.

SECONDARY OUTCOMES:
Algometry for assessing pressure pain thresholds (Pain sensitivity) | pre-intervention (T0), and inmmediate post-intervention (T1) (between the first and the second measurement, about 60 minutes have elapsed because it is done on the same day)
  An algometer shall be used to assess pain thresholds to pressure, i.e. squeezing so that pressure is converted into pain at two points. One point in the symphysis pubis area, and one point near the tibial tuberosity
maximal pelvic floor muscle strength (measured in grams and with the phenix device) | pre-intervention (T0), and inmmediate post-intervention (T1) (between the first and the second measurement, about 60 minutes have elapsed because it is done on the same day)
  Three measurements of maximal pelvic floor strength shall be performed with an intracavitary probe and the mean of the three measurements of maximal pelvic floor muscle strength shall be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Ferran Cuenca Martínez, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided